CLINICAL TRIAL: NCT02178332
Title: Yhteispeli: Intervention Effectiveness on Elementary School Childrens' Socio-emotional Skills and Psychiatric Symptoms
Brief Title: Yhteispeli - Effectiveness Study on Promoting Childrens' Socio-emotional Skills in School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Olli Kiviruusu, Research Manager, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THL/455/6.00.00/2014
Record Dates: First submitted 2014-04-03; First posted 2014-06-30 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Children's Socio-emotional Skills and Psychiatric Symptoms
Keywords: Children; socio-emotional; socio-emotional skills; psychiatric symptoms; SDQ; Finland; School; School community; Teacher; Whole school approach; Intervention; Effectiveness study; Cluster randomised trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yhteispeli, whole school programme (Experimental): Yhteispeli-programme aims to support children's socio-emotional skills and well being at schools. Schools receive the Yhteispeli manual and teachers receive 3 and head masters 2 lecture days about use of Yhteispeli methods including group discussions and exercises. In addition every school is visited 4 times to support the use of Yhteispeli methods. (Lectures for the head masters March 2013 - November 2013, teachers August 2013 - January 2014)
  Interventions: Other: Yhteispeli, whole school programme
- Two theoretical lectures (Active Comparator): Teachers receive two theoretical lectures on development of children's socio-emotional skills (3 hours in November 2013 and 3 hours in March 2014 ).
  Interventions: Other: Two theoretical lectures

INTERVENTIONS:
Other: Yhteispeli, whole school programme
  Arms: Yhteispeli, whole school programme
Other: Two theoretical lectures
  Arms: Two theoretical lectures

SUMMARY:
The purpose of this cluster randomised trial is to investigate whether the Yhteispeli whole school programme is effective in improving children's socio-emotional skills and mental health and socio-emotional skills.

All Finnish elementary schools and their classes in 1-3 grades were invited to participate in the study. The schools were randomly allocated to receive either Yhteispeli programme or two lectures

ELIGIBILITY:
Inclusion Criteria:

* All children from volunteering elementary schools and classes (grades 1 to 3) whose parents gave consent to participate

Exclusion Criteria:

* None

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4400 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Change in children's psychiatric symptoms | 6 months after baseline and 18 months after baseline
  SDQ - The Strengths and Difficulties Questionnaires
Change in children's socio-emotional skills | 6 months after baseline and 18 months after baseline
  A set of socio-emotional skills tests A set of questions regarding bullying

SECONDARY OUTCOMES:
Change in children's emotion recognition (and processing) | 6 months after baseline and 18 months after baseline
  A set of emotion recognition (and processing) tests
Change in children's executive functions | 6 months after baseline and 18 months after baseline
  A set of cognitive functions tests
Change in teacher and work community (occupational) wellbeing | 6 months after baseline and 18 months after baseline
  A set of teacher's occupational and work community wellbeing tests

OTHER OUTCOMES:
Change in teacher and parent interaction | 6 months after baseline and 18 months after baseline
  A set of teacher-parent interaction tests
Change in children's and teachers' perceptions of class environment | 6 months after baseline and 18 months after baseline
  A set of class environment questions rated by the teacher and children
Change in teaching and parenting styles | 6 months after baseline and 18 months after baseline
  A set of questions regarding child rearing
Change in teachers' and parents' socio-emotional skills | 6 months after baseline and 18 months after baseline
  A set of questions regarding adult socio-emotional skills

CONTACTS AND LOCATIONS:
Overall Officials: Olli Kiviruusu, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Olli Kiviruusu, Helsinki, Finland

REFERENCES:
- [Background] Bjorklund K, Liski A, Samposalo H, Lindblom J, Hella J, Huhtinen H, Ojala T, Alasuvanto P, Koskinen HL, Kiviruusu O, Hemminki E, Punamaki RL, Sund R, Solantaus T, Santalahti P. "Together at school"--a school-based intervention program to promote socio-emotional skills and mental health in children: study protocol for a cluster randomized controlled trial. BMC Public Health. 2014 Oct 7;14:1042. doi: 10.1186/1471-2458-14-1042. PMID 25287298
- [Result] Kiviruusu O, Bjorklund K, Koskinen HL, Liski A, Lindblom J, Kuoppamaki H, Alasuvanto P, Ojala T, Samposalo H, Harmes N, Hemminki E, Punamaki RL, Sund R, Santalahti P. Short-term effects of the "Together at School" intervention program on children's socio-emotional skills: a cluster randomized controlled trial. BMC Psychol. 2016 May 26;4(1):27. doi: 10.1186/s40359-016-0133-4. PMID 27230903